CLINICAL TRIAL: NCT04313296
Title: Prediction and Maintenance of Sinus Rhythm Among Atrial Fibrillation Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff shortage
Sponsor: Crystal Blake-Parlin (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Crystal Blake-Parlin, Program Supervisor-Lead Cardiac Ultrasound Sonographer, MaineHealth
Organization: MaineHealth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Blake-ParlinTOMTEC
Record Dates: First submitted 2019-01-29; First posted 2020-03-18 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a retrospective and prospective cohort study of patients with atrial fibrillation (AF) identified at Pen Bay Medical Center (PBMC). Patients will be identified for inclusion in the study based on a previous documented diagnosis of AF, have a documented echocardiogram, and have undergone electrical cardioversion, with a study enrollment goal of 150 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients identified at PBMC with a documented diagnosis of AF (Experimental): Patients identified at PBMC with a documented diagnosis of AF (at any point in time) and who have undergone any cardioversion.
  Interventions: Device: Unique measurement (AutoSTRAIN) by a commercial software program (TOMTEC-ARENA)

INTERVENTIONS:
Device: Unique measurement (AutoSTRAIN) by a commercial software program (TOMTEC-ARENA) — The historic echocardiograms from patients who meet the study inclusion criteria will be uploaded into this software, which was newly acquired by the PBMC Cardiology Department. MaineHealth Information Services are currently working with study staff to assure appropriate security compliance within the network. LA GLS has not been routinely collected previously from echocardiograms performed at PBMC because of a lack of such technology.

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disorder seen in clinical practice, with an estimated 2.7-6.1 million people in the U.S. affected by the disorder [1]. Previous studies have demonstrated that left atrial volume is a predictive measure of incident atrial fibrillation [2]. This study aims to add to the literature by investigating predictive measures of left atrial global longitudinal strain (LA GLS) that would be suggestive of maintenance of normal sinus rhythm post cardioversion. If the investigators could gain insight on the connection between LA GLS and cardioversion among patients with atrial fibrillation, the investigators could potentially help the clinical management of patients pre/post cardioversion, and potentially change poor outcomes.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a heart rhythm disorder in which the normal beating in the upper chambers of the heart is irregular, leading to poor blood flow to the lower chambers. Risk factors include older age, high blood pressure, obesity, European ancestry, diabetes, heart failure, ischemic heart disease, hyperthyroidism, chronic kidney disease, heavy alcohol use, and enlarged heart chambers on the left side [3]. AF increases a person's risk for stroke and contributes to an estimated 130,000 deaths each year [1]. Treatment generally includes medication, surgery, and/or healthy lifestyle changes [1]. Electrical cardioversion, in which the patient must undergo sedation or general anesthesia, is also used to convert patients with persistent AF to normal sinus rhythm. Electrical cardioversion has been associated with a high initial success rate of 68-98% [4], but long-term maintenance of sinus rhythm has proved challenging [5]. Due to the potential risks incurred to the patient, it is important to understand which patients are good candidates for cardioversion therapy. A review article describes that duration of AF, sex, age, weight smoking status, number of shocks at cardioversion, post-ablation procedure, medications, hypertension, diabetes, Chronic Obstructive Pulmonary Disease (COPD), obstructive sleep apnea, renal impairment, hyperthyroidism, coronary artery disease, congestive heart failure, left systolic dysfunction, left diastolic dysfunction, left ventricular hypertrophy, valvular heart disease, and left atrial size have each been found to be associated with maintenance of sinus rhythm [6].

Echocardiography has been increasing used in understanding the cardiac structure and risk of stroke among patients with AF, with left atrial size, left ventricular wall thickness, and left ventricular dysfunction recognized as independent predictors of AF [7]. Increasing evidence supports that the left atrial strain measurements can be a predictor of outcomes among AF patients, including stroke and AF recurrence after catheter ablation [8], [9]. The investigators aim to further explore left atrial strain measurements, including left atrial global longitudinal strain (LA GLS), as predictors of maintenance of normal sinus rhythm post- cardioversion. It is anticipated that a lower LA GLS will predict AF recurrence. To do this, the investigators will study patients with AF at Pen Bay Medical Center who have undergone cardioversion, measuring their LA GLS pre-cardioversion, and assess maintenance of sinus rhythm 6 months post-cardioversion. It is anticipated that this study will confirm LA GLS as a marker for maintenance of sinus rhythm post-cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* • Patients identified at PBMC with a documented diagnosis of AF (at any point in time) and who have undergone any cardioversion.

  * The patient would also need to have had an echocardiogram within six months pre-cardioversion (performed for any reason) with a well visualized atrial roof in order to perform the measurements accurately using the TOMTEC-ARENA software.

Exclusion Criteria:

* • Patients with a mitral regurgitation greater than moderate (effective regurgitant orifice >= .2 mm2)

  * Patients with post-surgical valve repair or replacement, if the procedure was done with a thoracotomy
  * Any patient how has had any cardiac surgery requiring a thoracotomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Blake-Parlin, Principal Investigator — Pen Bay Medical Center
Locations (1):
- Pen Bay Medical Center, Rockport, Maine, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Identified at PBMC(Pen Bay Medical Center) With a Documented Diagnosis of AF: Patients identified at PBMC with a documented diagnosis of AF (Atrial Fibrillation) (at any point in time) and who have undergone any cardioversion.
  Unique measurement (AutoSTRAIN) by a commercial software program (TOMTEC-ARENA): The historic echocardiograms from patients who meet the study inclusion criteria will be uploaded into this software, which was newly acquired by the PBMC Cardiology Department. MaineHealth Information Services are currently working with study staff to assure appropriate security compliance within the network. LA GLS has not been routinely collected previously from echocardiograms performed at PBMC because of a lack of such technology.
Period: Overall Study
Arm/Group | Patients Identified at PBMC(Pen Bay Medical Center) With a Documented Diagnosis of AF
Started | 209
Completed | 209
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Identified at PBMC With a Documented Diagnosis of AF
Number analyzed (Participants) | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 207
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 209
Patients Identified at PBMC with a documented diagnosis of AF [Count of Participants; unit: Participants] | 209

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Relationship Between Left Atrial Global Longitudinal Strain and the Maintenance of Sinus Rhythm After Cardioversion
Description: Left atrial global longitudinal strain as measured utilizing the TOMTECH - ARENA software program compared to duration of the maintenance of sinus rhythm following elective cardioversion.
  Time, in months, sinus rhythm was maintained.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Patients Identified at PBMC Who Underwent Cardioversion With a Diagnosis of AF: Patients identified at PBMC with a documented diagnosis of AF (at any point in time) and who have undergone any cardioversion.
  Unique measurement (AutoSTRAIN) by a commercial software program (TOMTEC-ARENA): The historic echocardiograms from patients who meet the study inclusion criteria will be uploaded into this software, which was newly acquired by the PBMC Cardiology Department. MaineHealth Information Services are currently working with study staff to assure appropriate security compliance within the network. LA GLS has not been routinely collected previously from echocardiograms performed at PBMC because of a lack of such technology.
Arm/Group | Patients Identified at PBMC Who Underwent Cardioversion With a Diagnosis of AF
Number analyzed (Participants) | 209
participants
  Maintained SR for >6 months | 85
  Did not maintain SR for 6 months | 124

ADVERSE EVENTS:
Time Frame: Adverse events were not collected as this study was a chart review. There were no interventions.
Description: This was a chart review. Most of the charts reviewed were retrospective. 26 subjects were prospective. Informed consent was obtained for the chart review. There were no interventions.
Arm/Group | Patients Identified at PBMC With a Documented Diagnosis of AF
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT04313296/Prot_SAP_000.pdf